CLINICAL TRIAL: NCT04163692
Title: Effects of Progressive Relaxation Training on Artralgia, Quality of Life and Emotional Status in Breast Cancer Patients Receiving Aromatatase Inhibitor Therapy
Brief Title: Progressive Relaxation Training in Breast Cancer Patients Receiving Aromatatase Inhibitor Therapy
Acronym: PREBCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Umut Bahçacı, Principal investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PREBCA
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Relaxation therapy; Pain; Aromatase Inhibitors
MeSH Terms: conditions — Breast Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: A computer generated list of random sequence numbers was created with 1:1 allocation ratio to randomise participants into study or control groups. Randomisation sequence was concealed until assignment of interventions. The group allocation was made by study researcher who implemented the PRE.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Progressive relaxation exercises (PRE) as 1 day supervised and 3 days home based program in a week, for 6 weeks
  Interventions: Other: Progressive relaxation exercises
- Control Group (No Intervention): Information was provided about pain and its treatment and the importance of relaxing exercises without any intervention, up to 6 weeks.

INTERVENTIONS:
Other: Progressive relaxation exercises — Following intructions have been performed by patients:
  * Punch your hands and contract your forearm
  * Punch your hands, push your elbow towards the seat
  * Bend your elbows
  * Push your shoulders back
  * Press your knee down and pull your toes towards you
  * Pull your knees towards you and push your feet down
  * Tighten your hips
  * Push your head back
  * Lift your eyebrows
  * Make wrinkles on your nose
  * Tighten your teeth
  * Push your chin down
  * Close your eyes and think of good things.
  Arms: Exercise Group

SUMMARY:
This study evaluates the effects of progressive relaxation exercises on artralgia, quality of life and anxiety-deppression in breast cancer patients receiving aromatase inhibitor. Half of the participants will receive supervised progressive relaxing exercises, while other half will not receive any exercise but only advice about relaxing.

Hypothesis: Progressive relaxation exercises improve the pain, quality of life and emotional status in breast cancer patients receiving aromatase inhibitor therapy.

DETAILED DESCRIPTION:
Aromatase inhibitors (AI) can cause musculoskeletal problems and increased risk of fracture as side effects in breast cancer (BC) survivors. In particular, arthralgia can be observed in almost 50% of patients receiving AI. Moreover; cognitive dysfunctions , decreases in quality of life , anxiety and depression , sleep problems and fatigue can be seen in some of patients receiving AI. According to these possible side effects, evaluation and treatment of such health profiles, pain and symptoms is important in terms of improving the quality of life of the patients.

Progressive muscle relaxation exercises (PRE) were first described by Jacobson in 1938. PRE are in use today with different arrangements and updates. It was well defined physiological, perceptual and behavioral positive findings of muscle relaxation.

PRE was thought to be effective on artralgia, quality of life and anxiety-depression in BC survivors receiving AI.

The patients have been searched from the medical records of brest health center in a local hospital. Necessary permissions to use this data was provided from medical coordinator of the hospital and from the coordinator of Breast Health Center.

The study was conducted as two armed, assessor blinded and randomised controlled trial. BC survivors who are receiving AI were randomised to study (performed PRE) or control (no intervention) group. Eligible patients were provided information about the the study and invited to participate in study via phone call. All assessments and exercise training was carried out in Physiotherapy Department of the same hospital. Outcomes were assessed baseline and at 6th-week intervention Primary endpoint was pain assessment assessed by Brief Pain inventory. Secondary endpoints were quality of life assessed by Functional Assessment of Chronic Illness Therapy and emotional status by Hospital Anxiety and Depression scales.

Statistical analysis Sample size was calculated by using a previous study mentioned the impact of yoga on functional outcomes in breast cancer survivors with aromatase inhibitor-associated arthralgias. The mean and standart deviation data of the FACT-B parameter was used with the power (1-type II error) of 0.80 and a type I error of 0.05. Therefore, it was aimed to recruit at least 20 participants per group. In total, with dropout rate of 30%, it was estimated to recruit 26 patients in each group.

Mean [95% confidence intervals (CI)], standard deviations and frequency rates was analyzed for baseline charecteristics. Group distributions were examined with the Kolmogorov Simirnov test. Groups analysis were performed using the non parametric test methods due to the low number of participants. Mann-Whitney U test for the analysis of quantitative independent data, and Wilcoxon test was used for the analysis of dependent data. Mc-Nemar Test was used for dependent variables and Chi-Square test was used for independent variables in the analysis of qualitative data. Cohen's Formula used for calculating efect size of differences between and within the groups. Figures are performed by the SPSS graphics. P value <0.05 was considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Using Aromatase Inhibitors for more than 6 months
* Diagnosis of breast cancer stage 1-3
* Postmenopausal woman aged under 70 years and with hormone-receptor positive
* Approval of physician for participating in PRE program

Exclusion Criteria:

* Participation on a regular physical training in the previous 6 months period
* Communication problems
* Neurological or ortopedical problems
* Presence of lyphedema diagnosis

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Brief pain inventory (BPI) | 24 hours
  Assesses the severity of pain and its impact on functioning. Consisting of 17 questions, evaluating pain location, severity, and pain status, especially in the last 24 hours. Scores of 3-4 are defined as mild, 5-7 as moderate, 8-10 as severe pain in this scale.

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy - Breast (FACT-B) | 7 days
  Evaluates the multidimensionel quality of life in patients with breast cancer and is available in many languages . The questionnaire includes 5 sub-scales that assess physical, social, emotional, functional and other anxiety status. It has 27-item general and 10-item breast cancer specific scale in which patients evaluate their status. Patients determine an appropriate expression for themselves in the last 7 days, with a 5 point scale as 0: none, 1: very little, 2: slightly, 3: quite, 4: too much. Higher scores indicate higher quality of life
Hospital Anxiety and Depression scale (HAD) | 7 days
  Consists of 14 questions which 7 of them evaluate depression and 7 of them evaluate anxiety. The cut-off score is 10/11 for the anxiety subscale and 7/8 for the depression subscale

CONTACTS AND LOCATIONS:
Overall Officials: Umut Bahcacı, MSc, Principal Investigator — Florence Nightingale Hospital, Istanbul; Zeynep Erdoğan İyigün, Asst. Prof., Principal Investigator — Florence Nightingale Hospital, Istanbul; Songul Atasavun Uysal, Prof., Principal Investigator — Hacettepe University; Çetin Ordu, Asst. Prof., Principal Investigator — Florence Nightingale Hospital, Istanbul; Vahit Özmen, Prof., Study Chair — Florence Nightingale Hospital, Istanbul; Gürsel Remzi Soybir, Prof., Study Chair — Memorial Etiler Health Center
Locations (1):
- Florence Nightingale Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a recent plan to make IPD available

REFERENCES:
- [Background] Cuzick J, Sestak I, Forbes JF, Dowsett M, Knox J, Cawthorn S, Saunders C, Roche N, Mansel RE, von Minckwitz G, Bonanni B, Palva T, Howell A; IBIS-II investigators. Anastrozole for prevention of breast cancer in high-risk postmenopausal women (IBIS-II): an international, double-blind, randomised placebo-controlled trial. Lancet. 2014 Mar 22;383(9922):1041-8. doi: 10.1016/S0140-6736(13)62292-8. Epub 2013 Dec 12. PMID 24333009
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Aromatase inhibitors versus tamoxifen in early breast cancer: patient-level meta-analysis of the randomised trials. Lancet. 2015 Oct 3;386(10001):1341-1352. doi: 10.1016/S0140-6736(15)61074-1. Epub 2015 Jul 23. PMID 26211827
- [Background] Mincey BA, Duh MS, Thomas SK, Moyneur E, Marynchencko M, Boyce SP, Mallett D, Perez EA. Risk of cancer treatment-associated bone loss and fractures among women with breast cancer receiving aromatase inhibitors. Clin Breast Cancer. 2006 Jun;7(2):127-32. doi: 10.3816/CBC.2006.n.021. PMID 16800971
- [Background] Bender CM, Sereika SM, Brufsky AM, Ryan CM, Vogel VG, Rastogi P, Cohen SM, Casillo FE, Berga SL. Memory impairments with adjuvant anastrozole versus tamoxifen in women with early-stage breast cancer. Menopause. 2007 Nov-Dec;14(6):995-8. doi: 10.1097/gme.0b013e318148b28b. PMID 17898668
- [Background] Cella D, Fallowfield L, Barker P, Cuzick J, Locker G, Howell A; ATAC Trialistsa9 Group. Quality of life of postmenopausal women in the ATAC ("Arimidex", tamoxifen, alone or in combination) trial after completion of 5 years' adjuvant treatment for early breast cancer. Breast Cancer Res Treat. 2006 Dec;100(3):273-84. doi: 10.1007/s10549-006-9260-6. Epub 2006 Jun 21. PMID 16944295
- [Background] Breckenridge LM, Bruns GL, Todd BL, Feuerstein M. Cognitive limitations associated with tamoxifen and aromatase inhibitors in employed breast cancer survivors. Psychooncology. 2012 Jan;21(1):43-53. doi: 10.1002/pon.1860. Epub 2010 Oct 21. PMID 20967847
- [Background] So WK, Marsh G, Ling WM, Leung FY, Lo JC, Yeung M, Li GK. The symptom cluster of fatigue, pain, anxiety, and depression and the effect on the quality of life of women receiving treatment for breast cancer: a multicenter study. Oncol Nurs Forum. 2009 Jul;36(4):E205-14. doi: 10.1188/09.ONF.E205-E214. PMID 19581224
- See also: incidence of breast cancer — http://gco.iarc.fr/today/data/factsheets/cancers/20-Breast-fact-sheet.pdf.